CLINICAL TRIAL: NCT05584735
Title: Determining the Relationship Between Gut Microbiota and Immune Response to Influenza or COVID-19 Vaccine in Immunosuppressed Patients With Inflammatory Bowel Disease
Brief Title: Determining the Relationship Between Gut Microbiota and Immune Response to Influenza or COVID-19 Vaccine
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0977; A534250 (Other: UW Madison); SMPH/MEDICINE/GASTROENT (Other: UW Madison); Protocol version 7/18/2024 (Other: UW Madison)
Record Dates: First submitted 2022-10-14; First posted 2022-10-18 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Crohn's disease; ulcerative colitis
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative | interventions — Influenza Vaccines; COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Saliva, and Fecal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants with Inflammatory Bowel Disease (IBD): Participants with IBD who are receiving a flu or COVID-19 vaccine
  Interventions: Biological: Influenza vaccine; Biological: COVID-19 vaccine

INTERVENTIONS:
Biological: Influenza vaccine — Observe effects of flu vaccine on microbiome
Biological: COVID-19 vaccine — Observe effects of COVID-19 vaccine on microbiome

SUMMARY:
This study will evaluate the effect of the microorganisms in the gut on how well the flu or COVID-19 vaccine works in people who have a weakened immune system due to inflammatory bowel disease. Participants can expect to be in the study for up to 65 days.

DETAILED DESCRIPTION:
The overall objective of this study is to evaluate the role of gut microbiome in influenza or COVID-19 vaccine response in immunosuppressed populations. Microbial diversity (alpha diversity) is decreased in immunosuppressed patients and might be associated with lower immunogenicity to vaccines.

It is known that patients with IBD have dysbiosis of their gut microbiome and those immunosuppressed may have a lower vaccine response. In this aim, the investigators will evaluate whether differences in microbial diversity predict immune response to the influenza and COVID-19 vaccine.

In this prospective study, immunosuppressed IBD patients will be vaccinated per standard of care and blood will be collected to measure the immune response. A fecal and saliva sample will be collected to characterize the gut microbiome. The investigators hypothesize that reduced richness / alpha-diversity in gut microbiota will correlate with those with a blunted vaccine response.

ELIGIBILITY:
Inclusion Criteria:

* A history of chronic (greater than 3 month) ulcerative colitis or Crohn's disease diagnosed and documented by the standard clinical, radiographic, endoscopic, and histopathologic criteria
* Currently one of the following groups:

  1. Group A: Anti-TNF Therapy Group

     * Maintenance monotherapy: infliximab (at least every 8 weeks), golimumab (at least monthly), adalimumab (at least every 2 weeks), or certolizumab (at least monthly)
     * Combination Therapy: Anti-TNF Combination Therapy Group on anti-TNF therapy as described above along with either methotrexate, azathioprine, or 6MP
  2. Group B: Non-TNG biologic

     * Ustekinumab Therapy: on either ustekinumab monotherapy or combination therapy with methotrexate, azathioprine, or 6MP
     * Vedolizumab Therapy: on either vedolizumab monotherapy or combination therapy with methotrexate, azathioprine, or 6MP
     * Risankizumab Therapy: 360mg at least every 8 weeks
  3. Group C: Janus Kinase Therapy

     * Tofacitinib Therapy: at least 5mg PO BID
     * Upadactinib Therapy: at least 15mg PO daily
* Patient has been on stable treatment for IBD for at least three months
* Must be able to provide research samples between 28-65 days post influenza or Covid-19 vaccination.

Exclusion Criteria:

* Member of a vulnerable group (pregnant, lacking consent capacity, non-English speaking)
* Recent oral antibiotics within previous 2 months

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants diagnosed with IBD
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2023-11-03 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Influenza or COVID-17 antibody concentrations | Baseline
  Hemagglutination inhibition assay (HIA) will be used to measure influenza antibodies in blood. COVID-19 antibody concentration analysis will be completed with LabCorp's Cov2Quant IgG™ assay which uses immunoassay that uses electrochemiluminescent technology (ECL) for quantitative determination of anti-receptor binding domain (RBD) IgG antibodies specific to SARS-CoV-2.
Influenza or COVID-19 antibody concentrations | One blood draw between 28-65 days after baseline
  Hemagglutination inhibition assay (HIA) will be used to measure influenza antibodies in blood. COVID-19 antibody concentration analysis will be completed with LabCorp's Cov2Quant IgG™ assay which uses immunoassay that uses electrochemiluminescent technology (ECL) for quantitative determination of anti-receptor binding domain (RBD) IgG antibodies specific to SARS-CoV-2.
Microbiome metrics | One stool collection between days 0-65
  Microbiome metrics will include phylogenetic diversity, and analyses of relative abundance of microbes using 16SrRNA gene sequence data from fecal material. Alpha diversity of the microbiome will be evaluated.
Microbiome stability | One stool collection between days 0-65
  Microbiome stability will be evaluated using hierarchical clustering of weighted and unweighted UniFrac distances (a beta diversity metric indexing compositional similarity/difference) for microbiome using 16SrRNA gene sequence data from fecal material.

SECONDARY OUTCOMES:
Correlation between Fecal Metabolomic Activity and Vaccine Response | up to 65 days
Correlation between Saliva DNA and Vaccine Response | up to 65 days

CONTACTS AND LOCATIONS:
Overall Officials: Freddy Caldera, DO, MS, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No